CLINICAL TRIAL: NCT06623591
Title: Ameliorating Effects and Mechanisms of Transcutaneous Auricular Vagus Nerve Stimulation on Constipation in Parkinson's Disease Patients: a Randomized, Double-blind Clinical Trial
Brief Title: Ameliorating Effects and Mechanisms of TaVNS on Constipation in PD Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kezhong Zhang (Other)
Responsible Party: Sponsor-Investigator, Kezhong Zhang, Professor, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-taVNS
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease, Idiopathic; Constipation
Keywords: constipation; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Transcutaneous auricular vagus nerve stimulation (Experimental): For Experimental Arm, active transcutaneous auricular vagus nerve stimulation, Patients underwent 28 consecutive daily sessions of taVNS.
  Interventions: Device: active Transcutaneous auricular vagus nerve stimulation
- Sham Transcutaneous auricular vagus nerve stimulation (Sham Comparator): For sham transcutaneous auricular vagus nerve stimulation arm, Sham Comparator, patients underwent 28 consecutive daily sessions of sham-taVNS (the electrodes were fixed at the the left earlobe).
  Interventions: Device: sham Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: active Transcutaneous auricular vagus nerve stimulation — Transcutaneous auricular vagus nerve stimulation was conducted by transcutaneous electrical stimulation therapy instrument to the cymba conchae of left ear in the vicinity of the auricular branch vagus nerve. Stimulation parameters: frequency = 20 Hz; pulse width = 500 μs, twice a day, 30 minutes each time.
  Arms: Active Transcutaneous auricular vagus nerve stimulation
Device: sham Transcutaneous auricular vagus nerve stimulation — In the sham stimulation group, the electrodes were fixed at the left earlobe with the same stimulus parameters. Stimulation parameters: frequency = 20 Hz; pulse width = 500 μs, twice a day, 30 minutes each time.
  Arms: Sham Transcutaneous auricular vagus nerve stimulation

SUMMARY:
The investigators intend to conduct a randomized, double-blind, sham-stimulation-controlled experiment, incorporating various clinical scales, gastrointestinal electrogram, and high-resolution anorectal manometry (HRAM), to investigate the improvement effect of taVNS on constipation symptoms in PD patients.

DETAILED DESCRIPTION:
The investigators intend to conduct a randomized, double-blind, sham-stimulation-controlled experiment, incorporating various clinical scales, gastrointestinal electrogram, and high-resolution anorectal manometry (HRAM), to investigate the improvement effect of taVNS on constipation symptoms in PD patients. Meanwhile, the investigators aimed to verify mechanistic effects by investigating changes in proteins and cytokines related to inflammation and intestinal barrier function in serum and feces to verify mechanistic effects.

ELIGIBILITY:
Inclusion Criteria:

1. aged 40-70 years;
2. had a PD diagnosis designated by movement disorder neurologists (Ke-zhong Zhang and Yong-sheng Yuan) according to Movement Disorder Society Clinical Diagnostic Criteria;
3. fulfilled Rome IV criteria for functional constipation, including having < 3 spontaneous bowel movements (SBM; i.e., not induced by rescue medication) per week for the past 3 months with symptom duration of at least 6 months;
4. stable initiation of PD medications, leastways 3 month before this investigation; (5) provided written informed consent.

Exclusion Criteria:

1. a history of previous abdominal surgery (other than appendectomy);
2. the presence of carcinoma;
3. any organic diseases causing constipation or neurologic diseases such as multiple sclerosis, rachischisis, or spinal cord injury;
4. taking antidepressant agents including tricyclic antidepressants and selective serotonin reuptake inhibitors;
5. a serious concomitant disease of the heart, liver, kidney, or diabetes;
6. pregnancy or lactation;
7. participating in another trial or enrolled in a trial during the past month;
8. an allergic reaction to surface electrodes.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
alterations in complete spontaneous bowel movements per week (CSBMs/week) | Assessed at 2 weeks before baseline, 2 weeks before the last day of intervention
  By having patients record their bowel movements two weeks before the start of the experiment and two weeks before the end of the experiment, calculate the CSBMs/week.

SECONDARY OUTCOMES:
Change from Baseline Gastrointestinal Dysfunction Scale for Parkinson's Disease (GIDS-PD) at one day post intervention | Assessed at baseline, one day post intervention
  The Gastrointestinal Dysfunction Scale for Parkinson's Disease is a novel disease-specific self-report tool to quantitatively assess the presence and severity of gastrointestinal dysfunction features in patients with PD, with strong reliability and validity. The GIDS-PD (Appendix S1) is a Likert self-report scale composed of 12 items. The total score of the GIDS-PD is computed by adding the total score of items 1 through 12, resulting in a minimum score of 1 and a maximum score of 108.
Change from Baseline Gastrointestinal Symptoms Rating Scales at one day post intervention | Assessed at baseline, one day post intervention
  Used to evaluate the gastrointestinal symptoms and discomfort level of patients, from 0 to 105.
Change from Baseline constipation symptoms scores at one day post intervention | Assessed at baseline, one day post intervention
  Used to evaluate the constipation symptoms , from 0 to 30.
Change from Baseline Patient Assessment of Constipation Quality of Life scale，PAC-QOL at one day post intervention | Assessed at baseline, one day post intervention
  Used to evaluate quality of life, a total of 28 items are divided into 4 aspects: physiological discomfort, psychological discomfort, palpitations, and satisfaction. The PAC-QOL score range is 0-4, with lower scores indicating better results.
Change from Baseline Patient Assessment of Constipation Symptoms questionnaire at one day post intervention | Assessed at baseline, one day post intervention
  Used to evaluate the constipation symptoms , from 0 to 48.
Change from Baseline HRAM at one day post intervention--Resting pressure (mmHg) | Assessed at baseline, one day post intervention
  Following HRV test, HRAM was undertaken using a solid-state manometric instrument with 12 circumferential sensors spaced at 1 cm intervals and an outer diameter of 4.2 mm to evaluate anorectal sensorimotor function. Patients were asked to be in the left lateral position with the hips and knees flexed, and then the solid-state catheter was inserted into the rectum through the anal orifice. After a 3-minute period of stabilization, the sequential maneuver procedures are as follows: Resting pressure (mmHg), maximum squeeze pressure (mmHg). First-sensation volume, desire to defecate threshold, and maximum tolerance were tested by constant dilation of balloon
Change from Baseline HRAM at one day post intervention--maximum squeeze pressure (mmHg) | Assessed at baseline, one day post intervention
  Following HRV test, HRAM was undertaken using a solid-state manometric instrument with 12 circumferential sensors spaced at 1 cm intervals and an outer diameter of 4.2 mm to evaluate anorectal sensorimotor function. Patients were asked to be in the left lateral position with the hips and knees flexed, and then the solid-state catheter was inserted into the rectum through the anal orifice. After a 3-minute period of stabilization, the sequential maneuver procedures are as follows: Resting pressure (mmHg), maximum squeeze pressure (mmHg). First-sensation volume, desire to defecate threshold, and maximum tolerance were tested by constant dilation of balloon
Change from Baseline HRAM at one day post intervention--First sensation (mL) | Assessed at baseline, one day post intervention
  Following HRV test, HRAM was undertaken using a solid-state manometric instrument with 12 circumferential sensors spaced at 1 cm intervals and an outer diameter of 4.2 mm to evaluate anorectal sensorimotor function. Patients were asked to be in the left lateral position with the hips and knees flexed, and then the solid-state catheter was inserted into the rectum through the anal orifice. After a 3-minute period of stabilization, the sequential maneuver procedures are as follows: Resting pressure (mmHg), maximum squeeze pressure (mmHg). First-sensation volume, desire to defecate threshold, and maximum tolerance were tested by constant dilation of balloon
Change from Baseline HRAM at one day post intervention--desire to defecate threshold | Assessed at baseline, one day post intervention
  Following HRV test, HRAM was undertaken using a solid-state manometric instrument with 12 circumferential sensors spaced at 1 cm intervals and an outer diameter of 4.2 mm to evaluate anorectal sensorimotor function. Patients were asked to be in the left lateral position with the hips and knees flexed, and then the solid-state catheter was inserted into the rectum through the anal orifice. After a 3-minute period of stabilization, the sequential maneuver procedures are as follows: Resting pressure (mmHg), maximum squeeze pressure (mmHg). First-sensation volume, desire to defecate threshold, and maximum tolerance were tested by constant dilation of balloon
Change from Baseline HRAM at one day post intervention--maximum tolerance | Assessed at baseline, one day post intervention
  Following HRV test, HRAM was undertaken using a solid-state manometric instrument with 12 circumferential sensors spaced at 1 cm intervals and an outer diameter of 4.2 mm to evaluate anorectal sensorimotor function. Patients were asked to be in the left lateral position with the hips and knees flexed, and then the solid-state catheter was inserted into the rectum through the anal orifice. After a 3-minute period of stabilization, the sequential maneuver procedures are as follows: Resting pressure (mmHg), maximum squeeze pressure (mmHg). First-sensation volume, desire to defecate threshold, and maximum tolerance were tested by constant dilation of balloon
Change from Baseline gastrointestinal electrogram at one day post intervention--amplitude | Assessed at baseline, one day post intervention
  A total of 8 leads cover the body surface projection of the stomach and intestines, which can reflect the gastrointestinal motility
Change from Baseline gastrointestinal electrogram at one day post intervention--frequency | Assessed at baseline, one day post intervention
  A total of 8 leads cover the body surface projection of the stomach and intestines, which can reflect the gastrointestinal motility.
Change from Baseline serum indicators at one day post intervention | Assessed at baseline, one day post intervention
  A blood sample was taken at 8 a.m. at baseline and after 4 weeks of treatment. For each patient, about 5 mL of blood was drawn into a procoagulant tube and 4 mL into 2 anticoagulant tubes with EDTA; it was centrifuged at 4°C and 1139g for 10 minutes and 5 minutes respectively. The serum in the procoagulant tube was divided into 3 portions, and the plasma in the anticoagulant tubes was divided into 2 portions - each about 0.5 mL - and placed at -80°C for assay within 6 months.
Change from Baseline feces indicators at one day post intervention | Assessed at baseline, one day post intervention
  placed at -80°C for assay within 6 months.
Change from Baseline The motor part of the Unified Parkinson's Disease Rating Scale at one day post intervention | Assessed at baseline, one day post intervention
  The measure mainly reflects the overall severity of Parkinson's disease motor symptoms. The minimum and maximum values of the motor part of the Unified Parkinson's Disease Rating Scale are 0 and 108. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No